CLINICAL TRIAL: NCT04841278
Title: Utility of Combined EUS and ERCP Procedures in the Evaluation of Liver Graft Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decided not to go ahead with study
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5170383
Record Dates: First submitted 2017-10-28; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Liver Graft Dysfunction

STUDY DESIGN:
Intervention Model Description: Single prospective arm with historical controls as comparator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EUS/ERCP (Experimental): Patients with liver graft dysfunction enrolled sequentially for proposed protocol: EUS with possible interventions and possible ERCP
  Interventions: Device: EUS/ERCP

INTERVENTIONS:
Device: EUS/ERCP — EUS with possible interventions, including liver biopsy and/or cholangiography, and possible ERCP. No new experimental procedures are proposed, only new protocol for diagnosis and treatment of liver graft dysfunction.

SUMMARY:
The purpose of this investigator-initiated study is to determine whether a single-step session that combines endoscopic ultrasound (which may further include liver biopsy and needle-guided cholangiography) with endoscopic cholangiopancreatography (ERCP) can facilitate in the management of liver graft dysfunction. All patients will undergo the same procedural protocol.

DETAILED DESCRIPTION:
Liver graft dysfunction can arise from many disease processes, which include biliary obstruction, rejection, infection and ischemia. Battery of tests, and at times empiric therapy, is necessary to obtain final diagnosis. This results in waste of time and medical resources that can lead to delay in care, which may ultimately translate to increase morbidity and mortality, as well as increase in cost.

In this protocol, the investigators propose utilization of interventional endoscopy for the diagnosis and treatment of liver graft dysfunction. Use of endoscopic ultrasound (EUS) with possible liver biopsy and cholangiography, and endoscopic retrograde cholangiopancreatography in one session may facilitate diagnosis and treatment. All patients enrolled in this protocol will undergo the same procedural protocol. The quality of care metrics in these patients (such as length of stay, cost, mortality, etc), will be compared to that of historical controls.

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized patients with liver graft dysfunction

Exclusion Criteria:

* Thrombocytopenia (platelets <50.000/mL) until corrected
* Coagulopathy (international normalized ratio (INR) >1.5) until corrrected
* Use of thrombolytic or anti-platelet agents within 5-7 days of the procedure.
* Any with known bleeding diathesis will be excluded. (e.g. disseminated intravascular coagulation (DIC), von-Willebrand disease, hemophilia).
* Those who had recent prior liver biopsy or EUS/ERCP will be excluded.
* Those with active bacteremia will be excluded, at least until treated.
* For this initial study, those with altered GI tract anatomy (e.g. those with hepaticojejunostomy or gastro-jejunostomy) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to final diagnosis | Up to 30 days
  Time from first diagnostic test to final diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Alexander W Jahng, MD, Principal Investigator — Loma Linda University

IPD SHARING:
Plan to Share IPD: No